CLINICAL TRIAL: NCT05176600
Title: Pilot Study on the Evaluation of the Functionality, Safety and Feasibility of a Bimanual Robotic Exoskeletal Platform for the Treatment of the Upper Limb in Patients With Stroke
Brief Title: Bimanual Robotic Exoskeletal Platform for the Treatment of the Upper Limb in Patients With Stroke. A Feasibility Study
Acronym: Birehab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wearable Robotics srl. (Industry)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Lucia Lencioni, CEO, Wearable Robotics srl.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDG_Birehab_2021
Record Dates: First submitted 2021-11-10; First posted 2022-01-04 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bimanual group (Experimental): In this group, patients will perform a robotic rehabilitation based on bimanual serious games
  Interventions: Device: Robotic rehabilitation using the Arm Light Exoskeleton Rehab Station (ALEx RS) and bimanual serious games
- Unimanual group (Active Comparator): In this group, patients will perform a robotic rehabilitation based on unimanual serious games
  Interventions: Device: Robotic rehabilitation using the Arm Light Exoskeleton Rehab Station (ALEx RS) and unimanual serious games

INTERVENTIONS:
Device: Robotic rehabilitation using the Arm Light Exoskeleton Rehab Station (ALEx RS) and bimanual serious games — Patients will undergo a bimanual 30-session robotic rehabilitation, using the robot ALEx RS with the bimanual configuration and the related serious games. Each session will last 45 minute. Daily sessions will be provided, five days a week.
  Arms: Bimanual group
Device: Robotic rehabilitation using the Arm Light Exoskeleton Rehab Station (ALEx RS) and unimanual serious games — Patients will undergo a unimanual 30-session robotic rehabilitation, using the robot ALEx RS with the unimanual configuration and the related serious games.Daily sessions will be provided, five days a week.
  Arms: Unimanual group

SUMMARY:
The purpose of the study is to test the technical functionality, safety, and feasibility of a bimanual robotic exoskeletal platform and associated serious games in order to offer information on technological and functional advances that will be included in the device's finalization.

In addition, a secondary goal will be to assess the therapeutic effects of a rehabilitation therapy based on the bimanual configuration, comparing it to a unimanual treatment delivered on the same platform (using the specific configuration).

ELIGIBILITY:
Inclusion Criteria:

* height between 150 and 190 cm;
* weight not exceeding 130 kg;
* ischemic injury;
* first cortical and supra-tentorial event;
* moderate motor deficit of the upper limb (score on the Fugl-Meyer Assessment - Upper Extremity between 29 and 42);
* time since stroke event between 1 and 6 months;
* trunk control test score greater than or equal to 48;
* healthy bone density and skeleton that does not suffer from unhealed fractures.

Exclusion Criteria:

* Relevant medical comorbidities (severe neurological diseases, cardiovascular diseases, diabetes / unstabilized hypertension);
* Cognitive impairment that prevents understanding of the exercises administered;
* Unavailability to provide informed consent;
* Pregnant women;
* Severe spasticity (Ashworth 4);
* Major muscle contractures;
* Excessive asymmetry in the length of the arms;
* Upper limb prostheses;
* Excessive joint limitations that make it difficult or painful to use the device;
* Use of pacemakers or implantation of active devices;
* Patients who already participate in another clinical study or who are already undergoing another similar robotic rehabilitation treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and description | through the study, an average of 10 months
  Number and description of adverse events related to the provided intervention

SECONDARY OUTCOMES:
Changes in EEG-based Interhemispheric coupling index | Before the intervention, after a 1-hour robotic rehabilitation session
  Interhemispheric coupling evaluated by means of 64-channel Electroencephalogram (EEG)
Changes in EEG-based Interhemispheric coupling index | Before the intervention, after a 6-week robotic rehabilitation intervention
  Interhemispheric coupling evaluated by means of 64-channel Electroencephalogram (EEG)
Changes in EEG-based Interhemispheric coupling index | Before the intervention, 1 week after the end of the 30-session robotic intervention
  Interhemispheric coupling evaluated by means of 64-channel Electroencephalogram (EEG)
Changes in EEG-based Connectivity index | Before the intervention, after a 1-hour robotic rehabilitation session
  Connectivity evaluated by means of 64-channel Electroencephalogram (EEG)
Changes in EEG-based Connectivity index | Before the intervention, after a 6-week robotic rehabilitation intervention
  Connectivity evaluated by means of 64-channel Electroencephalogram (EEG)
Changes in EEG-based Connectivity index | Before the intervention, 1 week after the end of the 30-session robotic intervention
  Connectivity evaluated by means of 64-channel Electroencephalogram (EEG)
Changes in Fugl-meyer Assessment Upper Extremity motor functioning | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a stroke-specific, performance-based impairment index. It ranges from 0 (hemiplegia) to 66 points (normal).
Changes in Fugl-meyer Assessment - Sensory functioning | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a stroke-specific, sensory impairment index. It ranges from 0 (worse) to 12points (best).
Changes in Modified Ashworth Scale | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a validated measure of spasticity. It ranges from 0 (normal) to 4 (rigid limb).
Changes in Motricity Index for upper extremity | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a validated measure of upper limb strength. It ranges from 0 (worse) to 100 (normal strength).
Changes in Wolf Motor Function Test | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a validated measure of upper extremity motor ability through timed and functional tasks.
  The scores ranges from 0 to 75; lower scores are indicative of lower functioning levels.
Changes in Action Research Arm Test (ARAT) | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a valid measure of upper-extremity functional limitation. The total score on the ARAT ranges from 0 to 57, with the lowest score indicating that no movements can be performed, and the upper score indicating normal performance.
Changes in Execution time (seconds) measured with the robot | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is the time (in seconds) required to perform reaching movement using the robot
Changes in Range of Motion (degrees) measured with the robot | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is the range of motion (measured in degrees) of shoulder and elbow evaluated using the robot
Changes in Number of velocity peaks measured with the robot | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a measure of movement smoothness while performing reaching movements with the robot.
System Usability Scale | After a 6-week robotic rehabilitation intervention
  It is a self-administered questionnaire to evaluate usability. It ranges from 0 to 100. Higher scores mean better usability.
Technology Acceptance Model (TAM) | After a 6-week robotic rehabilitation intervention
  It is a self-administered questionnaire to evaluate the acceptance of the provided.
  It comprises several questions rated on a 7-point likert scale.
Likert for Satisfaction | After a 6-week robotic rehabilitation intervention
  Satisfaction will be assessed using a 11-point likert scale. It ranges from 0 to 10. Higher scores mean higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Aprile, MD, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (1):
- Fondazione Don Carlo Gnocchi, Rome, Italy

REFERENCES:
- [Derived] Mauro MC, Fasano A, Germanotta M, Cortellini L, Insalaco S, Pavan A, Comanducci A, Guglielmelli E, Aprile IG. Aperiodic brain activity changes in patients with stroke following virtual reality-based upper limb robotic rehabilitation: a pilot Randomized Controlled Trial. Front Hum Neurosci. 2025 Oct 17;19:1671804. doi: 10.3389/fnhum.2025.1671804. eCollection 2025. PMID 41179260